CLINICAL TRIAL: NCT02223754
Title: Evaluation of an Investigational Multifocal Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-5593
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lotrafilcon B / etafilcon A (Active Comparator): Subject randomized to this sequence will first be dispensed the lotrafilcon B contact lens and then the etafilcon A contact lens.
  Interventions: Device: lotrafilcon B; Device: etafilcon A
- etafilcon A / lotrafilcon B (Experimental): Subject randomized to this sequence will first be dispensed the etafilcon A contact lens and then the lotrafilcon B contact lens.
  Interventions: Device: lotrafilcon B; Device: etafilcon A

INTERVENTIONS:
Device: lotrafilcon B — Soft contact lens to be worn as daily wear, monthly replacement modality.
  Other Names: AirOptix Aqua Multifocal
Device: etafilcon A — Soft contact lens to be worn as daily wear, daily disposable modality.

SUMMARY:
The purpose of this study is to test the performance of an investigational multifocal test soft contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were required to have read, understand, and signed the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Between 40 and 70 years of age.
4. Subjects must own a wearable pair of spectacles, if required for their distance vision.
5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration)
6. Already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire"*
7. The subject's vertex corrected spherical equivalent distance refraction was required to be in the range +3.50 to -5.75 in each eye.
8. Refractive cylinder ≤ -0.75 D in each eye.
9. ADD power in the range +0.75 D to +2.50 D in each eye.
10. Best corrected visual acuity of 20/20-3 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who became pregnant during the study were discontinued).
2. Any ocular or systemic allergies that may have contraindicated contact lens wear.
3. Any ocular or systemic disease, autoimmune disease, or use of medication, that may have contraindicated contact lens wear.
4. Any ocular abnormality that may have interfered with contact lens wear.
5. Use of any ocular medication, with the exception of rewetting drops.
6. Any previous intraocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
7. History of herpetic keratitis.
8. History of binocular vision abnormality or strabismus.
9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV).
10. History of diabetes.
11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
12. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which may contraindicate contact lens wear.
13. Any ocular infection or inflammation.
14. Any corneal distortion or irregular cornea.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Montgomery, Alabama
  - Mission Viejo, California
  - Jacksonville, Florida
  - Orange Park, Florida
  - Saint Augustine, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Pittsburg, Kansas
  - East Lansing, Michigan
  - Vestal, New York
  - Denver, North Carolina
  - Powell, Ohio
  - Springfield, Ohio
  - Warwick, Rhode Island
  - Memphis, Tennessee
  - Tyler, Texas
  - Salem, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled a total of 371 subjects. Of those enrolled subjects 49 did not meet the eligibility criteria and 322 subjects were dispensed a study lens. Of the dispensed subjects 297 completed the study and 25 were discontinued from the study.
Groups:
- Etafilcon A / Lotrafilcon B: Subjects were randomized to one of two lens sequences. Subjects first received the etafilcon A contact lens and then received the Control lens (lotrafilcon B contact lens.
- Lotrafilcon B/ Etafilcon A: Subjects were randomized to one of two lens sequences. Subjects first received the lotrafilcon B lens and then received the etafilcon A lens.
Period: Period 1
Arm/Group | Etafilcon A / Lotrafilcon B | Lotrafilcon B/ Etafilcon A
Started | 163 | 159
Completed | 159 | 144
Not Completed | 4 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Test Article No Longer Available | 1 | 5
Not completed — Unsatisfactory Visual Response | 0 | 1
Period: Period 2
Arm/Group | Etafilcon A / Lotrafilcon B | Lotrafilcon B/ Etafilcon A
Started | 159 | 144
Completed | 156 | 141
Not Completed | 3 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lens Discomfort | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Test Article No Longer Available | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population consists of subjects that were dispensed a study lens.
Groups:
- Etafilcon A / Lotrafilcon B; Lotrafilcon B / Etafilcon A: Subjects that were randomized to this sequence and were dispensed a study lens.
- Total: Total of all reporting groups
Arm/Group | Etafilcon A / Lotrafilcon B | Lotrafilcon B / Etafilcon A | Total
Number analyzed (Participants) | 163 | 159 | 322
Age, Continuous [Mean (Standard Deviation); unit: years]
  Hyperopes, N=59, N=53, N=112 | 52.3 (6.59) | 51.9 (7.04) | 52.1 (6.78)
  Myopes, N=104, N=106, N=210 | 49.3 (6.10) | 49.5 (5.77) | 49.4 (5.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 120 | 248
  Male | 35 | 39 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Black or African American | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 147 | 144 | 291
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 163 | 159 | 322

OUTCOME MEASURES:

1. Primary Outcome: Overall Quality of Vision Using the Contact Lens User Experience (CLUE) TM Questionnaire
Description: CLUE Overall Quality of Vision is assessed using the Contact Lens User Experience (CLUE)TM questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 8 -12 days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A: Subjects that received the etafilcon A contact lens during either the first or second period of the study.
- Lotrafilcon B: Subjects that received the lotrafilcon B contact lens during either the first or second period of the study.
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
units on a scale
  Hyperopes, N=94, N=94 | 51.15 (21.647) | 54.28 (20.749)
  Myopes, N=181, N=181 | 53.55 (18.644) | 51.84 (19.319)

2. Primary Outcome: Distance Binocular Visual Acuity (LogMAR)
Description: Distance time controlled LogMAR Visual Acuity was carried out binocularly with high luminance and high contrast.
Time Frame: 8- 12 Days post wear
Population: The analysis population consists of subjects that have completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Lotrafilcon B: Subjects that received the lotrafilcon B during either the first or second period of the study.
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
LogMAR
  Hyperopes, N=94, N=94 | -0.069 (0.0908) | -0.066 (0.0982)
  Myopes, N=180, N=181 | -0.100 (0.0991) | -0.093 (0.0981)

3. Primary Outcome: Intermediate Binocular Visual Acuity (LogMAR)
Description: Intermediate time controlled LogMAR Visual Acuity was carried out binocularly using High lumiance and High Contrast.
Time Frame: 8-12 days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
LogMAR
  Hyperopes, N=94, N=94 | -0.061 (0.0829) | -0.050 (0.0897)
  Myopes, N=180, N=181 | -0.081 (0.0803) | -0.063 (0.0894)

4. Primary Outcome: Near Binocular Visual Acuity (LogMAR)
Description: Near time controlled LogMAR Visual Acuity was carried out binocularly using High lumiance and High Contrast.
Time Frame: 8-12 days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
LogMAR
  Hyperopes, N=94, N=94 | 0.050 (0.0970) | 0.074 (0.1035)
  Myopes, N=180, N=181 | 0.034 (0.1039) | 0.049 (0.1176)

5. Primary Outcome: Corneal Staining
Description: Corneal staining is evaluated using Sodium Fluorescein strips. The Fluorescien strip was lightly placed on the subject's inferior palpebral conjunctiva. The corneal Staining was graded using the scale Grade 0: No Staining, Grade 1: Trace(Minimal superficial staining or stippling), Grade 2: Mild (Regional or diffuse punctate staining), Grade 3:Moderate(Significant dense coalesced staining, corneal abrasion or foreign body tracks.), Grade 4 Severe(Severe abrasions greater than 2 mm in diameter, ulcerations, epithelial loss, or full thickness abrasion.). The data was dichotomized into two group subjects with grade 3 or higher staining, and those subjects with less than Grade 3. Below the percentage of subject eyes with grade 3 or higher is reported for each lens.
Time Frame: 8 - 12 Days post wear
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation. The analysis was conducted on subject eyes.
Measure: Number; unit: percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
Number analyzed (Subject Eyes) | 550 | 550
percentage of Subject Eyes
  Hyperopes, N=188, N=188 | 0.0 | 0.0
  Myopes, N=362, N=362 | 0.0 | 0.0

6. Primary Outcome: Bulbar Conjunctival Injection
Description: The bulbar is the scelra. Bulbar Conjunctival Injection was assessed using an Efron Grading scale by 1 unit increments. Grade 0: Normal, Grade 1: Trace, Grade 2: Mild, Grade 3: Moderate, Grade 4:Severe. The data was dichotomized into two group subjects with grade 3 or higher Conjunctival injection, and those subjects with less than Grade 3. Below the percentage of subject eyes with grade 3 or higher is reported for each lens.
Time Frame: 8- 12 Days post wear
Population: as for outcome 5
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
Number analyzed (Subject Eyes) | 550 | 550
Percentage of Subject Eyes
  Hyperopes, N=188, N=188 | 0.0 | 0.0
  Myopes, N=362 , N=362 | 0.0 | 0.0

7. Primary Outcome: Limbal Conjunctival Injection
Description: The Limbus is the 1 to 2mm wide zone of conjunctiva and underlying tissue adjacent to where the cornea joins the sclera. Limbal Conjunctival Injection was assesed using the Efron grading scale in 1 unit increments. Grade 0: Normal, Grade 1: Trace, Grade 2: Mild, Grade 3: Moderate, Grade 4:Severe. The data was dichotomized into two group subjects with grade 3 or higher Conjunctival injection, and those subjects with less than Grade 3. Below the percentage of subject eyes with grade 3 or higher is reported for each lens.
Time Frame: 8- 12 Days post wear
Population: as for outcome 5
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
Number analyzed (Subject Eyes) | 550 | 550
Percentage of Subject Eyes
  Hyperopes, N=188, N=188 | 0.0 | 0.0
  Myopes, N=362, N=362 | 0.0 | 0.0

8. Primary Outcome: Contact Lens Fitting
Description: Contact Lens fitting is reported as a binary response. Yes- acceptable lens fit, No- unacceptable lens fit. The percentage of subject eyes with acceptable fit is reported.
Time Frame: 8- 12 Days post wear
Population: as for outcome 5
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Etafilcon A | Lotrafilcon B
Number analyzed (Participants) | 275 | 275
Number analyzed (Subject Eyes) | 550 | 550
Percentage of Subject Eyes
  Hyperopes, N=188, N=188 | 100 | 100
  Myopes, N=362, N=362 | 99.5 | 100

ADVERSE EVENTS:
Time Frame: Approximately 8-12 days per intervention.
Arm/Group | Etafilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/307 | 0/318
Other Adverse Events (participants affected / at risk) | 0/307 | 0/318

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days